CLINICAL TRIAL: NCT02561884
Title: A Single-dose, Randomized, Two-period, Two-treatment, Two-sequence, Crossover Bioequivalence Study on a Olostar Tab Versus Two Co-administered Reference Products Olmesartan Medoxomil and Rosuvastatin Calcium in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DW_DWJ1276006
Record Dates: First submitted 2015-09-24; First posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AB (Experimental): Olostar Tab. followed by Olmetec and Crestor
  Interventions: Drug: Olostar Tab.; Drug: Co-administration of Olmetec and Crestor
- BA (Experimental): Olmetec and Crestor followed by Olostar Tab.
  Interventions: Drug: Olostar Tab.; Drug: Co-administration of Olmetec and Crestor

INTERVENTIONS:
Drug: Olostar Tab.
Drug: Co-administration of Olmetec and Crestor

SUMMARY:
To demonstrate the bioequivalence of a Olostar Tab versus two co-administered reference IMPs Olmetec and Crestor.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 18.5 and ≤ 30.0 kg/m2.
* No clinically significant findings in a 12-lead electrocardiogram (ECG)
* Age 18-60 years at screening

Exclusion Criteria:

* History of severe allergy or allergic reactions to the IMPs or related drugs
* History of serious clinical illness that can impact fate of drugs including major surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
AUC | 0~72hr
Cmax | 0~72hr